CLINICAL TRIAL: NCT03252457
Title: A Multicenter Prospective Randomized Study of Dexamethasone Combined With Decitabine Versus Dexamethasone in the Treatment of Newly Diagnosed Primary Immune Thrombocytopenia (ITP)
Brief Title: Decitabine Combining Dexamethasone Versus Dexamethasone in Management of ITP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Collaborators: Second Affiliated Hospital of Medical College Shandong University (Other); Shandong Provincial Hospital (Other Government); Qingdao Central Hospital (Other); Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAC in ITP
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic; Immune Thrombocytopenia
Keywords: Purpura; Thrombocytopenia; immune throbocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Purpura; Thrombocytopenia | interventions — Decitabine; Dexamethasone; Hydrocortisone

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- combination treatment group (Experimental): 100 enrolled patients are randomly picked up to take decitabine in combination with dexamethasone at the indicated dose
  Interventions: Drug: Decitabine; Drug: Dexamethasone
- single treatment group (Active Comparator): 100 enrolled patients are randomly picked up to take dexamethasone at the indicated dose
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Decitabine — given intravenously at a dose of 3.5mg/m2/d for 4 consecutive days as a cycle and repeated every 2 weeks for 3cycles
  Other Names: pharmachemie
  Arms: combination treatment group
Drug: Dexamethasone — given 40mg/d for 4 consecutive days as a cycle , If platelet count remained below 30 × 109/L or there were bleeding symptoms by day 10, an additional cycle of dexamethasone was given.
  Other Names: Hydrocortisone

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University and other 18 well-known hospitals in China. In order to report the efficacy and safety of decitabine combining with dexamethasone for the treatment of adults with immune thrombocytopenia (ITP), compared to dexamethasone alone .

DETAILED DESCRIPTION:
The investigators anticipate to undertaking a parallel group, multicentre, randomised controlled trial of 200 ITP adult patients from 19 medical centers in China. One part of the participants are randomly selected to receive dexamethasone (given 40mg/d for 4 consecutive days as a cycle , If platelet count remained below 30 × 109/L or there were bleeding symptoms by day 10, an additional cycle of dexamethasone was given) combining with decitabine (given intravenously at a dose of 3.5mg/m2/d for 4 consecutive days as a cycle and repeated every 2 weeks for 3 cycles), the others are selected to receive dexamethasone therapy(given 40mg/d for 4 consecutive days as a cycle, If platelet count remained below 30 × 109/L or there were bleeding symptoms by day 10, an additional cycle of dexamethasone was given). Platelet count, bleeding and other symptoms were evaluated before and after treatment, adverse events are also recorded throughout the study in order to report the efficacy and safety of the combination therapy compared to dexemathasone alone therapy for the treatment of adults with ITP.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for immune thrombocytopenia.
2. within 3 months fromdiagnosis,untreated patients, may be male or female, between the ages of 18 ~ 80 years.
3. To show a platelet count < 30×10^9/L, and with bleeding manifestations.
4. Eastern Cooperative Oncology Group（ECOG）performance status ≤ 2.

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit.
2. Received high-dose steroids or intravenous immunoglobulin transfusion(IVIG) in the 3 weeks prior to the start of the study.
3. Current HIV infection or hepatitis B virus or hepatitis C virus infections.
4. Severe medical condition (lung, hepatic or renal disorder) other than ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)
5. Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period.
6. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.
7. Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of platelet response(continuous response rate) | up to 1 year per subject
  Complete Response:a sustained (≥ 3 months) platelet count ≥100×10^9/L;response: a sustained (≥ 3 months) platelet count ≥ 30×10^9/L without recurrence of thrombocytopenia;No response (NR): platelet count < 30 × 10^9/L or a less than two fold increase in platelet count from baseline or the presence of bleeding. Platelet count must be measured on two occasions more than a day apart.

SECONDARY OUTCOMES:
therapy associated adverse events | up to 1 year per subject
  The number and frequency of therapy associated adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, Dr, Principal Investigator — Shandong University
Locations (1):
- Qilu hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182
- [Result] Zhou H, Hou Y, Liu X, Qiu J, Feng Q, Wang Y, Zhang X, Min Y, Shao L, Liu X, Li G, Li L, Yang L, Xu S, Ni H, Peng J, Hou M. Low-dose decitabine promotes megakaryocyte maturation and platelet production in healthy controls and immune thrombocytopenia. Thromb Haemost. 2015 May;113(5):1021-34. doi: 10.1160/TH14-04-0342. Epub 2015 Jan 8. PMID 25566808
- [Result] Wei Y, Ji XB, Wang YW, Wang JX, Yang EQ, Wang ZC, Sang YQ, Bi ZM, Ren CA, Zhou F, Liu GQ, Peng J, Hou M. High-dose dexamethasone vs prednisone for treatment of adult immune thrombocytopenia: a prospective multicenter randomized trial. Blood. 2016 Jan 21;127(3):296-302; quiz 370. doi: 10.1182/blood-2015-07-659656. Epub 2015 Oct 19. PMID 26480931
- [Result] Din B, Wang X, Shi Y, Li Y. Long-term effect of high-dose dexamethasone with or without low-dose dexamethasone maintenance in untreated immune thrombocytopenia. Acta Haematol. 2015;133(1):124-8. doi: 10.1159/000362529. Epub 2014 Sep 20. PMID 25247485